CLINICAL TRIAL: NCT05382429
Title: Official Title:Observation of the Clinical Efficacy of Two Surgical Procedures on the Short-term Outcome of Moderate Varus Knee Osteoarthritis
Brief Title: Observation of the Clinical Efficacy of Two Surgical Procedures for Varus Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: chenjinli
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; high tibial osteotomy; medial collateral ligament; fracture healing
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Before initiating the trial, an investigator who was not involved in the study generated a computer-generated randomization list (block length 10, ratio 1:1). Allocation concealment was achieved by using opaque, sealed, sequentially numbered envelopes containing details of group assignment. Assignment occurred after baseline information was recorded. According to preoperative allocation, the patients were given open wedge high tibial osteotomy or closingwedge high tibial osteotomy.For the open wedge high tibial osteotomy group, Those who were randomly assigned to the OWHTO group, OWHTO Surgical procedure will be performed.For the closing wedge high tibial osteotomy group, hose who were randomly assigned to the CWHTO group, CWHTO Surgical procedure will be performed.
Who Masked: Outcomes Assessor
Masking Description: Whereas patients and surgeons were aware of the group assignments, the outcome assessors and data analysts were remained blinded during the study period.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OWHTO (Experimental): open wedge high tibial osteotomy group For the open wedge high tibial osteotomy group, Those who were randomly assigned to the OWHTO group, OWHTO Surgical procedure will be performed.
  Interventions: Procedure: OWHTO
- CWHTO (Experimental): closing wedge high tibial osteotomy group For the closing wedge high tibial osteotomy group, hose who were randomly assigned to the CWHTO group, CWHTO Surgical procedure will be performed
  Interventions: Procedure: CWHTO

INTERVENTIONS:
Procedure: OWHTO — OWHTO Surgical procedure For the OWHTO Surgical procedure, only medial split biplanar osteotomy performed.
  Arms: OWHTO
Procedure: CWHTO — CWHTO Surgical procedure For the OWHTO Surgical procedure, only lateral closure osteotomy was performed.
  Arms: CWHTO

SUMMARY:
The purpose of this study is to conduct a prospective randomized controlled trial to compare the effects between two surgical procedures in the treatment of varus knee osteoarthritis.The hypothesis was that there would be no difference in mechanical axis correction between two surgical procedures.

DETAILED DESCRIPTION:
This was a single-center, prospective, double-blinded, randomized controlled trial, comparing two surgical procedures in the treatment of varus knee osteoarthritis. Participants were recruited from September 2019 to September 2021. Before initiating the trial, an investigator who was not involved in the study generated a computer-generated randomization list (block length 10, ratio 1:1). Allocation concealment was achieved by using opaque, sealed, sequentially numbered envelopes containing details of group assignment. Assignment occurred after baseline information was recorded. Whereas participants and surgeons were aware of the group assignments, the outcome assessors and data analysts were remained blinded during the study period. Operations were performed by the same team of sports medicine surgeons under general anesthesia.For the open wedge high tibial osteotomy group, Those who were randomly assigned to the OWHTO group, OWHTO Surgical procedure will be performed. For the closing wedge high tibial osteotomy group, hose who were randomly assigned to the CWHTO group, CWHTO Surgical procedure will be performed. The sample size calculation was based on data from previous studies. Accepting an α risk of 0.05 and a β risk of 0.2 in a bilateral contrast, the minimum sample size required for each group was 35. To compensate for an estimated 15% loss to follow up, at least 82 patients would be included.

ELIGIBILITY:
Inclusion Criteria:

The eligibility criteria for HTO were spontaneous osteonecrosis of the knee of the medial femoral condyle, medial compartment OA, Ahlbäck grades 1 or 2, femorotibial angle (FTA) of ≤185, flexion contracture of ≤15° , lack of damage to the anterior cruciate ligament (ACL) and posterior cruciate ligament, and no age restrictions .

Exclusion Criteria:

Congenital deformity of knee joint, severe rheumatoid arthritis, Charkoff's joint, injury of knee joint (injury of medial and lateral collateral ligament, patella fracture, etc.) or surgical history (meniscectomy, femoral or tibial fracture after surgery), large number of free bodies or soft tissue flexion contracture in the joint >10º, and range of motion of knee joint <100º.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
The Visual Analog Scale score | Baseline
  Assess pain on a scale of 0 (no pain) to 10 (worst possible pain).
The Visual Analog Scale score | Postoperative 6 months
  Assess pain on a scale of 0 (no pain) to 10 (worst possible pain).
The Visual Analog Scale score | Postoperative 12 months
  Assess pain on a scale of 0 (no pain) to 10 (worst possible pain).
The Visual Analog Scale score | Postoperative 18 months
  Assess pain on a scale of 0 (no pain) to 10 (worst possible pain).
Radiological evaluation | Baseline
  Items include hip-knee-ankle (HKA), the medioproximal tibial angle(MPTA) and joint line Angle retraction(JLCA)
Radiological evaluation | Postoperative 6 months
  Items include hip-knee-ankle (HKA), the medioproximal tibial angle(MPTA) and joint line Angle retraction(JLCA)
Radiological evaluation | Postoperative 12 months
  Items include hip-knee-ankle (HKA), the medioproximal tibial angle(MPTA) and joint line Angle retraction(JLCA)
Radiological evaluation | Postoperative 18 months
  Items include hip-knee-ankle (HKA), the medioproximal tibial angle(MPTA) and joint line Angle retraction(JLCA)
WOMAC | Baseline
  This score evaluates the structure and function of the knee joint from three aspects of pain, stiffness and physical function, covering the basic symptoms and signs of the whole OA. The lower the score, the better the functional status of the patient.WOMAC score < 21 is mild, 21 to 48 is moderate, > 48 is classified as severe.
WOMAC | Postoperative 6 months
  This score evaluates the structure and function of the knee joint from three aspects of pain, stiffness and physical function, covering the basic symptoms and signs of the whole OA. The lower the score, the better the functional status of the patient.WOMAC score < 21 is mild, 21 to 48 is moderate, > 48 is classified as severe.
WOMAC | Postoperative 12 months
  This score evaluates the structure and function of the knee joint from three aspects of pain, stiffness and physical function, covering the basic symptoms and signs of the whole OA. The lower the score, the better the functional status of the patient.WOMAC score < 21 is mild, 21 to 48 is moderate, > 48 is classified as severe.
WOMAC | Postoperative 18 months
  This score evaluates the structure and function of the knee joint from three aspects of pain, stiffness and physical function, covering the basic symptoms and signs of the whole OA. The lower the score, the better the functional status of the patient.WOMAC score < 21 is mild, 21 to 48 is moderate, > 48 is classified as severe.
The hospital for surgery score | Baseline
  The clinical efficacy was evaluated by HSS knee function score. Items include pain, function, activity level, etc., with a total score of 0 to100, the higher the score, the better the curative effect.
The hospital for surgery score | Postoperative 6 months
  The clinical efficacy was evaluated by HSS knee function score. Items include pain, function, activity level, etc., with a total score of 0 to100, the higher the score, the better the curative effect.
The hospital for surgery score | Postoperative 12 months
  The clinical efficacy was evaluated by HSS knee function score. Items include pain, function, activity level, etc., with a total score of 0 to100, the higher the score, the better the curative effect.
The hospital for surgery score | Postoperative 18 months
  The clinical efficacy was evaluated by HSS knee function score. Items include pain, function, activity level, etc., with a total score of 0 to100, the higher the score, the better the curative effect.

SECONDARY OUTCOMES:
Postoperative complications | Postoperative 3 day
  Intraoperative blood loss, operation time, postoperative drainage, incidence of thrombosis, postoperative nerve damage
Postoperative complications | Postoperative 3 months
  Intraoperative blood loss, operation time, postoperative drainage, incidence of thrombosis, postoperative nerve damage

CONTACTS AND LOCATIONS:
Locations (1):
- Jinli Chen, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Proposals should be directed to lichunpu2020@163.com. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website .
URL: http://www.medresman.org.cn/uc/sindex.aspx